CLINICAL TRIAL: NCT06133270
Title: A Phase I, Randomised, Double Blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Once-daily Oral Doses of NNC0560-0004 in Healthy Humans, With an Additional Open Label Single Dose Cohort of CYP2D6 Poor Metabolizers.
Brief Title: A First Human Dose Study Investigating Safety and Concentration of Study Medicine in the Blood Following Once Daily Oral Dosing of NNC0560-0004 in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6561-7567; U1111-1285-1593 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers - Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0560-0004 (Experimental): The study will be conducted in 3 parts.
  Participants will be randomized to receive NNC0560-0004 in Part A: Single ascending dose (SAD) Part B: Multiple ascending dose (MAD)
  No randomisation - only active treatment in Part C: Single dose
  Interventions: Drug: NNC0560-0004
- Placebo (NNC0560-0004) (Placebo Comparator): Participant will be randomized to receive placebo in:
  Part A: Single ascending dose (SAD) Part B: Multiple ascending dose (MAD)
  Interventions: Drug: Placebo (NNC0560-0004)

INTERVENTIONS:
Drug: NNC0560-0004 — NNC0560-0004, Oral administration (taken through the mouth)
  Arms: NNC0560-0004
Drug: Placebo (NNC0560-0004) — Placebo matching NNC0560-0004, Oral administration (taken through the mouth)
  Arms: Placebo (NNC0560-0004)

SUMMARY:
In this trial, medicine NNC0560-0004 given in capsule form will be compared to placebo in healthy volunteers.

Participants will either get NNC0560-0004 or placebo. Which treatment they get is decided by chance.

This is a first in human trial, which means that this is the first time that NNC0560-0004 is given to humans.

The study will last for about two weeks plus the screening period (approximately 42 days) which in all is about 8 weeks.

Women must be of non-childbearing potential thus you cannot take part if you are pregnant, can become pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Key inclusion criteria:

1. Female, of non-childbearing potential, or male, both genders aged 18-55 years (both inclusive) at the time of signing informed consent.
2. Body Mass Index (BMI) between 18.5 and 29.9 kg/m^2 (both inclusive) at screening.
3. Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests including inflammatory markers performed during the screening visit, as judged by the investigator
4. CYP2D6 phenotype:

   1. For Part A and Part B: ultra-rapid (from cohort A3 forward and B1 forward), normal or intermediate CYP2D6 function
   2. For Part C: CYP2D6 Poor Metaboliser function

Key exclusion criteria:

1. Any disorder/condition, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
2. Known history of histamine intolerance or severe anaphylactic reactions
3. Abnormal values at screening for any of the following laboratory parameters

   * Aspartate aminotransferase (AST) greater than Upper limit of normal (ULN)+10%.
   * Alanine aminotransferase (ALT) greater than ULN +10%.
   * Bilirubin (except if known Gilbert's syndrome) greater than ULN +10%.
   * Creatinine greater than ULN.

     a.eGFR below 90 ml/min/1.73m^2
   * Glycated haemoglobin (HbA1c) greater than or equal to 5.7% (39 mmol/mol).
4. CYP2D6 unknown phenotype

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Part A: Number of treatment-emergent adverse events (TEAE) | From pre-dose (day 1) to end of study, Part A (up to day 13)
  Number of events
Part B: Number of treatment-emergent adverse events (TEAE) | From pre-dose (day 1) to end of study, Part B (up to day 26)
  Number of events
Part C: Number of treatment-emergent adverse events (TEAE) | From pre-dose (day 1) to end of study, Part C (up to day 84)
  Number of events

SECONDARY OUTCOMES:
Part A: AUC0-∞, SD: the area under the NNC0560-0004 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to end of study, Part A (up to day 13)
  h*nmol/L
Part A: Cmax, SD: the maximum plasma concentration of NNC0560-0004 after a single dose | From pre-dose (day 1) to end of study, Part A (up to day 13)
  nmol/L
Part A: tmax, SD: the time to maximum concentration of NNC0560-0004 after a single dose | From pre-dose (day 1) to end of study, Part A (up to day 13)
  hour
Part A:t½, SD: the terminal half-life of NNC0560-0004 after a single dose | From pre-dose (day 1) to end of study, Part A (up to day 13)
  hour
Part B: AUC0-24h, MD: the area under the NNC0560-0004 plasma concentration-time curve in the dosing interval after last dosing | From pre-dose on day 14 until end of study, Part B (up to day 26) (24 hours post-dose)
  h*nmol/L
Part B: Cmax, MD: the maximum plasma concentration of NNC0560-0004 after last dosing | From pre-dose on day 14 to end of study, Part B (up to day 26)
  nmol/L
Part B:tmax, MD: the time to maximum concentration of NNC0560-0004 after last dosing | From pre-dose on day 14 to end of study, Part B (up to day 26)
  hour
Part B:t½, MD: the terminal half-life of NNC0560-0004 after last dosing | From pre-dose on day 14 to end of study, Part B (up to day 26)
  hour
Part C: AUC0-∞, SD: the area under the NNC0560-0004 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to end of study, Part C (up to day 84)
  h*nmol/L
Part C: Cmax, SD: the maximum plasma concentration of NNC0560-0004 after a single dose | From pre-dose (day 1) to end of study, Part C (up to day 84)
  nmol/L
Part C: tmax, SD: the time to maximum concentration of NNC0560-0004 after a single dose | From pre-dose (day 1) to end of study, Part C (up to day 84)
  hour
Part C: t½, SD: the terminal half-life of NNC0560-0004 after a single dose | From pre-dose (day 1) to end of study, Part C (up to day 84)
  hour

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Northwick Park Hosptial, Watford, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com